CLINICAL TRIAL: NCT02482831
Title: The Difference in Duration of Sciatic Nerve Block Between Diabetic and Non-diabetic Patients
Acronym: DSNBD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Professor, Peking Union Medical College Hospital
Other Study IDs: anesthesiologyPUMCH002
Record Dates: First submitted 2015-06-15; First posted 2015-06-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Sciatic Nerve Block
Keywords: Sciatic nerve block; block duration; Semmes Weinstein monofilaments; fasting blood glucose; nerve block; sensory block duration; motor block duration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Diabetes: Diabatic participants who experienced unilateral lower limb surgery and received an ultrasound-guided (nerve stimulator assisted) subgluteal sciatic nerve block with 0.75% ropivacaine 20ml in Peking Union Medical College Hospital were selected.
  Interventions: Procedure: Subgluteal sciatic nerve block
- non-Diabetes: Non-diabatic participants who experienced unilateral lower limb surgery and received an ultrasound-guided (nerve stimulator assisted) subgluteal sciatic nerve block with 0.75% ropivacaine 20ml in Peking Union Medical College Hospital were selected.
  Interventions: Procedure: Subgluteal sciatic nerve block

INTERVENTIONS:
Procedure: Subgluteal sciatic nerve block — All patients (either diabetic or non-diabetic patients) received an ultrasound-guided (nerve stimulator assisted) subgluteal sciatic nerve block with 0.75% ropivacaine 20ml.

SUMMARY:
This study aims to compare the sensory and motor block duration and the incidence of nerve injury after sciatic nerve block between diabetic and non-diabetic patients, and screen for the factors that may affect the block recovery.

DETAILED DESCRIPTION:
This is an observational study. All participants who experienced unilateral lower limb surgery and received an ultrasound-guided (nerve stimulator assisted) subgluteal sciatic nerve block with 0.75% ropivacaine 20ml in Peking Union Medical College Hospital were selected. They were further assigned to either diabetic group or non-diabetic group according to their medical history (primary exposure). The primary end point was the sensory and motor block duration. These durations in terms of sensory and motor blocks of sciatic nerve(dorsal side, plantar side) were assessed at baseline, every 2 hours in 48 hours after the block (except for the second night). In addition, the associations between fasting blood glucose, glycosylated hemoglobin (hemoglobin A1c, HbA1c) and the degree of diabetic retinopathy and the durations of sensory and motor block were also examined. This is not a intervention study, because we will examine the outcomes between diabetic or non-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists :I-III;
* Age>=18 years;
* Undergo unilateral lower limb surgery;
* Sign consent form.

Exclusion Criteria:

* Refuse regional Anesthesia;
* Thresh of sensory >10g;
* Dyskinesia;
* Bleeding disorder;
* Regional skin infection;
* Regional drug allergy;
* Renal disfunction;
* Incompliant to study;
* Drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo unilateral lower limb surgery in Peking Union Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Duration of sensory block | 48 hours
  Sensory block is measured by Semmes Weinstein monofilaments. The block is measured at baseline, and every 2hours in 48 hours after the block.
Duration of motor block | 48 hours
  Motor blocks is visualized. The block is measured at baseline, and every 2hours in 48 hours after the block

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD, Principal Investigator — Peking Union Medical College University
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Gebhard RE, Nielsen KC, Pietrobon R, Missair A, Williams BA. Diabetes mellitus, independent of body mass index, is associated with a "higher success" rate for supraclavicular brachial plexus blocks. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):404-7. doi: 10.1097/AAP.0b013e3181ada58d. PMID 19920415
- [Background] Kalichman MW, Calcutt NA. Local anesthetic-induced conduction block and nerve fiber injury in streptozotocin-diabetic rats. Anesthesiology. 1992 Nov;77(5):941-7. doi: 10.1097/00000542-199211000-00017. PMID 1443749
- [Background] Kroin JS, Buvanendran A, Williams DK, Wagenaar B, Moric M, Tuman KJ, Kerns JM. Local anesthetic sciatic nerve block and nerve fiber damage in diabetic rats. Reg Anesth Pain Med. 2010 Jul-Aug;35(4):343-50. doi: 10.1097/aap.0b013e3181e82df0. PMID 20607875
- [Result] Cuvillon P, Reubrecht V, Zoric L, Lemoine L, Belin M, Ducombs O, Birenbaum A, Riou B, Langeron O. Comparison of subgluteal sciatic nerve block duration in type 2 diabetic and non-diabetic patients. Br J Anaesth. 2013 May;110(5):823-30. doi: 10.1093/bja/aes496. Epub 2013 Jan 24. PMID 23348203
- [Result] Sertoz N, Deniz MN, Ayanoglu HO. Relationship between glycosylated hemoglobin level and sciatic nerve block performance in diabetic patients. Foot Ankle Int. 2013 Jan;34(1):85-90. doi: 10.1177/1071100712460366. PMID 23386766
- [Result] Kroin JS, Buvanendran A, Tuman KJ, Kerns JM. Effect of acute versus continuous glycemic control on duration of local anesthetic sciatic nerve block in diabetic rats. Reg Anesth Pain Med. 2012 Nov-Dec;37(6):595-600. doi: 10.1097/AAP.0b013e31826742fd. PMID 22996200
- [Derived] Tang S, Wang J, Tian Y, Li X, Cui Q, Xu M, Song X, Zheng Y, Yang H, Ma C, Zhan L, Zhu C, Zhang Y, Yao M, Huang Y. Sex-dependent prolongation of sciatic nerve blockade in diabetes patients: a prospective cohort study. Reg Anesth Pain Med. 2019 Jul 12:rapm-2019-100609. doi: 10.1136/rapm-2019-100609. Online ahead of print. PMID 31302640